CLINICAL TRIAL: NCT07035691
Title: Plasma Biomarkers in Stratifying Patients Referred Via the Lower Gastro-intestinal (LGI) Suspected Cancer Two-week Wait (2WW) Pathway
Brief Title: New bioMarkers tO straTIfy cOlorectal caNcer Referrals
Acronym: MOTION
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 321809; WT 10042913 (Other: Queen Mary University of London)
Record Dates: First submitted 2025-06-11; First posted 2025-06-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Carcinoma; Polyp; Colorectal Adenoma
Keywords: Colorectal cancer; Cancer; Polyp; Adenoma; Cancer surveillance; Flag symptoms; Liquid biopsy; Progastrin; Circulating biomarkers; Biomarkers; Risk stratification; Early diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Neoplasms; Adenoma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected and plasma separated and frozen. Only plasma will be stored beyond the study under appropriate HTA approval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with flag symptoms referred via 2 week wait pathway to exclude colorectal cancer.: An additional blood sample for the study.

SUMMARY:
The goal of this observational study is to evaluate if a blood test for circulating progastrin (hPG80) and transposable elements (TEs) can accurately predict colorectal cancer (CRC) or polyps in adult patients referred to the 2-week wait (2WW) or Straight to Test (STT) pathways for suspected lower gastrointestinal cancer.

The main questions it aims to answer are:

Can plasma hPG80 levels accurately predict a diagnosis of CRC or polyps in patients undergoing standard 2WW investigations? Can transposable elements (TEs) in the plasma serve as predictive biomarkers for CRC diagnosis in these patients? What are the patient preferences for different diagnostic tests for CRC, particularly a blood-based test compared to more invasive methods?

Participants will:

Provide a 20ml blood sample during a routine hospital visit for their 2WW diagnostic test (e.g., colonoscopy, CT Colon).

Undergo standard clinical investigations as determined by their treating clinicians.

Have their final diagnosis (cancer, polyp, or normal) correlated with their plasma hPG80 levels.

For a subset of 100 participants (25 with confirmed CRC, 75 non-cancer), have their plasma analyzed for circulating signatures using RNAseq and DNAseq.

Complete an electronic post-study questionnaire to explore their preferences and experiences with different CRC diagnostic tests used within the 2WW pathway.

DETAILED DESCRIPTION:
Current Challenges in CRC Diagnosis Currently, the 2WW pathway for bowel symptoms typically involves a stool-based faecal immunochemical test (FIT) before referral. While the 2WW pathway is vital for expedited diagnosis, a systematic review from 2009 revealed that only 9.5% of patients referred with lower gastrointestinal (GI) symptoms through this pathway are ultimately diagnosed with cancer. This low positive predictive value places immense pressure on an already overstretched healthcare system, leading to unnecessary invasive investigations, increased costs, and prolonged patient anxiety. There's a clear need for more accurate and less invasive diagnostic tools to better stratify patients.

Progastrin (hPG80) as a Biomarker hPG80, a circulating blood biomarker, is a precursor to gastrin and has shown promise in detecting various GI cancers, including CRC. In healthy individuals, hPG80 is typically undetectable as it's converted to gastrin. However, elevated hPG80 levels can be found in the plasma of many patients with both early and advanced GI malignancies. Studies have shown an elevated hPG80 level in CRC subjects compared to those with benign polyps. This study will investigate whether plasma hPG80 levels can accurately predict CRC or polyps in 2WW patients and distinguish the absence of cancer based on PG levels.

Transposable Elements (TEs) as Biomarkers Transposable elements (TEs), which are mobile genetic elements, are also emerging as potential cancer biomarkers. Recent research has linked TEs to various cancers, including CRC. The Dr. Madapura's lab has shown that transposable element-derived RNA signatures can be superior predictors of diseases. This study will explore the role of TEs in predicting CRC diagnosis within the 2WW referral cohort. Specifically, it will identify and evaluate TEs in the plasma of these patients as potential predictive biomarkers. The analysis will involve RNA sequencing (RNAseq) and nanopore DNA sequencing (DNAseq) of plasma samples to look for transcript signatures and epigenetic modifications of DNA.

Study Design and Population This is a prospective, observational, cohort study conducted at Barts Health NHS Trust, initially focusing on the Royal London Hospital site. The study will recruit 582 adult patients referred via the 2WW or Straight to Test (STT) pathways for suspected lower GI cancer. Eligible patients will be aged over 18 years, have no history of inflammatory bowel disease, and have a performance status of ECOG 0-2 (or 3, pending clinical assessment). Patients with a family history of CRC are not excluded. Those with a documented familial type of CRC, untreated solid organ cancers, or who are not fit for standard investigations will be excluded.

Data Collection and Analysis Upon informed consent, a 20ml venous blood sample will be collected from participants at their first clinical appointment, usually during a routine hospital visit for their 2WW diagnostic test (e.g., colonoscopy, CT colonography). This sample will be used for both PG and TE analysis. Plasma PG levels will be measured, and a subset of 100 samples (25 confirmed CRC and 75 non-cancer samples) will undergo RNAseq and DNAseq for TE analysis.

The primary objective is to determine the sensitivity and specificity of plasma hPG80 levels in diagnosing CRC and benign colonic polyps. This will involve calculating positive and negative predictive values, and performing Receiver Operating Characteristic (ROC) curve analysis to assess the discriminatory ability of PG.

The secondary objective is exploratory and focuses on identifying and validating novel TEs as potential biomarkers for CRC diagnosis. This will involve the RNAseq and DNAseq analysis of the selected 100 samples.

A tertiary objective involves a post-study patient questionnaire survey to understand patient preferences and choices regarding CRC diagnostic tests, exploring their experience with a blood-based test compared to more invasive methods. This will be distributed electronically via SurveyMonkey™.

Expected Outcomes and Benefits

The study aims to provide crucial insights into whether adding a simple blood test (hPG80 and/or TE analysis) to the existing 2WW pathway can:

Improve diagnostic accuracy and speed: Leading to more effective and timely treatment.

Alleviate patient stress: By providing quicker and more accurate diagnoses, reducing anxiety associated with uncertainty.

Reduce unnecessary invasive procedures: Potentially avoiding colonoscopy-related complications and overall costs for the NHS.

Prioritize urgent cases: By better stratifying patients, allowing healthcare resources to be directed to those most in need.

There are no direct benefits to the study participants, but the knowledge gained is expected to have a significant long-term clinical impact on screening for suspected lower GI malignancies.

The study is funded by a research grant from LAPResearch UK.

ELIGIBILITY:
Inclusion Criteria:

* Adult, lower GI 2WW and or Straight to Test (STT) referral patients with suspected lower GI cancer.
* Male and Female patients aged >18 years.
* 2WW referral patients with no history of inflammatory bowel disease.
* Performance status (ECOG 0-2; and 3 pending clinical assessment of fitness).
* Patients with capacity to consent to the study.

Exclusion Criteria:

* Any patients referred outside of the 2WW and or STT referral pathways with suspected Lower GI cancer or those referred as an emergency with or suspected CRC.
* Age < 18 years.
* Patients not fit for standard investigations (e.g. not fit for gastroscopy, colonoscopy or CT colonography) in the 2WW pathway.
* Patients with no capacity to consent or who declined consent for participation.
* Patients with untreated solid organ cancers.
* Patients with known inflammatory bowel disease.
* Patients with documented familial type CRC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are referred by the GPs to the Barts Health NHS trust under the 2WW referral pathway and the STT pathway would be potentially eligible. We are planning to recruit patients initially only from the Royal London Hospital site and there is potential to expand recruitment to other hospital sites of Barts Health NHS Trust, if necessary.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of hPG80 to identify colorectal cancer and adenomatous polyp | From enrollment to 8 weeks (or until the 2WW diagnostic test is completed and the outcome available).
  Sensitivity and Specificity of hPG80 to determine colorectal cancer and adenomatous polyp
Identification of Transposable Element (TE) signatures in plasma of colorectal cancer patients | From enrollment to 8 weeks (or until the 2WW diagnostic test is completed and the outcome available).
  Expression of transposable element (TE) signatures in the plasma of patients with colorectal cancer and adenomatous polyps compared to healthy controls.

OTHER OUTCOMES:
Patient preference and choice of diagnostic tests for colorectal cancer | 12 weeks post recruitment date
  Survey based assessment of patient preferences and choices of different tests used in the colorectal 2WW pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Thaha, MBBS, FRCS, PhD, PGCe Hlt Econ, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD used in the publications might be shared under strict regulations.

REFERENCES:
- [Background] Reggiardo RE, Maroli SV, Peddu V, Davidson AE, Hill A, LaMontagne E, Aaraj YA, Jain M, Chan SY, Kim DH. Profiling of repetitive RNA sequences in the blood plasma of patients with cancer. Nat Biomed Eng. 2023 Dec;7(12):1627-1635. doi: 10.1038/s41551-023-01081-7. Epub 2023 Aug 31. PMID 37652985
- [Background] Alix-Panabieres C, Pantel K. Liquid Biopsy: From Discovery to Clinical Application. Cancer Discov. 2021 Apr;11(4):858-873. doi: 10.1158/2159-8290.CD-20-1311. PMID 33811121
- [Background] Lykoskoufis NMR, Planet E, Ongen H, Trono D, Dermitzakis ET. Transposable elements mediate genetic effects altering the expression of nearby genes in colorectal cancer. Nat Commun. 2024 Jan 25;15(1):749. doi: 10.1038/s41467-023-42405-0. PMID 38272908
- [Background] Prieur A, Cappellini M, Habif G, Lefranc MP, Mazard T, Morency E, Pascussi JM, Flaceliere M, Cahuzac N, Vire B, Dubuc B, Durochat A, Liaud P, Ollier J, Pfeiffer C, Poupeau S, Saywell V, Planque C, Assenat E, Bibeau F, Bourgaux JF, Pujol P, Sezeur A, Ychou M, Joubert D. Targeting the Wnt Pathway and Cancer Stem Cells with Anti-progastrin Humanized Antibodies as a Potential Treatment for K-RAS-Mutated Colorectal Cancer. Clin Cancer Res. 2017 Sep 1;23(17):5267-5280. doi: 10.1158/1078-0432.CCR-17-0533. Epub 2017 Jun 9. PMID 28600477
- [Background] You B, Mercier F, Assenat E, Langlois-Jacques C, Glehen O, Soule J, Payen L, Kepenekian V, Dupuy M, Belouin F, Morency E, Saywell V, Flaceliere M, Elies P, Liaud P, Mazard T, Maucort-Boulch D, Tan W, Vire B, Villeneuve L, Ychou M, Kohli M, Joubert D, Prieur A. The oncogenic and druggable hPG80 (Progastrin) is overexpressed in multiple cancers and detected in the blood of patients. EBioMedicine. 2020 Jan;51:102574. doi: 10.1016/j.ebiom.2019.11.035. Epub 2019 Dec 24. PMID 31877416

DOCUMENTS (2):
  • Study Protocol (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT07035691/Prot_000.pdf
  • Informed Consent Form (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT07035691/ICF_001.pdf